CLINICAL TRIAL: NCT06937073
Title: Comparative Study of Multi-component Real-time Remote Rehabilitation and Self Rehabilitation in the Treatment of Sarcopenia
Brief Title: Multi-component Real-time Remote Rehabilitation in Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Linbo Peng, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCHSCU-2024-2455
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; remote rehabilitation; muscle strength; real-time remote rehabilitation
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Single center, non blinded, randomized controlled, dual arm trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): In the "Fugu Medical" WeChat mini program, the intervention plan for the intervention group included: (1) dietary intake guidance and (2) exercise guidance. (1) Dietary intake guidance: The dietary guidance was mainly based on the general dietary guidelines for the elderly issued by the Chinese Nutrition Society. (2) Exercise guidance Exercise guidance included resistance training and balance training.
  Interventions: Behavioral: dietary intake guidance and exercise guidance
- Arm 2 (Active Comparator): Participants in the control group only received rehabilitation program articles in the form of images and text through the mobile application. These materials also included dietary intake guidance and exercise instructions. The frequency and intensity of the exercise instructions were sent to the patients at the same time. However, their daily adherence, including whether the training was completed or whether the dietary intake was appropriate, was not checked, verified, or followed up.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: dietary intake guidance and exercise guidance — In the "Fugu Medical" WeChat mini program, the intervention plan for the intervention group included: (1) dietary intake guidance and (2) exercise guidance.
  1. Dietary intake guidance: The dietary guidance was mainly based on the general dietary guidelines for the elderly issued by the Chinese Nutrition Society.
  2. Exercise guidance Exercise guidance included resistance training and balance training.
  Arms: Arm 1
Behavioral: Control — Participants in the control group only received rehabilitation program articles in the form of images and text through the mobile application. These materials also included dietary intake guidance and exercise instructions. The frequency and intensity of the exercise instructions were sent to the patients at the same time. However, their daily adherence, including whether the training was completed or whether the dietary intake was appropriate, was not checked, verified, or followed up.
  Arms: Arm 2

SUMMARY:
This study is designed as a single center, non blinded, randomized controlled, dual arm trial. We designed to allocate participants in a 1:1 ratio to compare the effects of real-time remote rehabilitation and self rehabilitation with multiple components on muscle strength, muscle mass, balance, and walking ability in patients with sarcopenia. Each participant signs an informed consent form before registering for the study. This protocol follows the 2013 Standard Protocol Project: Intervention Trial Recommendation Guidelines.

DETAILED DESCRIPTION:
This study is designed as a single center, non blinded, randomized controlled, dual arm trial. We designed to allocate participants in a 1:1 ratio to compare the effects of real-time remote rehabilitation and self rehabilitation with multiple components on muscle strength, muscle mass, balance, and walking ability in patients with sarcopenia. Each participant signs an informed consent form before registering for the study. This protocol follows the 2013 Standard Protocol Project: Intervention Trial Recommendation Guidelines.

ELIGIBILITY:
Inclusion Criteria:

According to the diagnostic criteria for sarcopenia established by the Asian Working Group for Sarcopenia (AWGS):

1. Low muscle strength:

   Handgrip strength < 28 kg for men, < 18 kg for women; and/or
2. Low physical performance:

   Usual gait speed (6-Meter Gait Speed, 6MGS) ≤ 1.0 m/s; and/or
3. Low muscle mass:

Skeletal Muscle Mass Index (SMI) < 7.0 kg/m² for men, < 5.7 kg/m² for women.

Exclusion Criteria:

1. Unable or unwilling to undergo body composition measurement.
2. Regular exercise habits within the past 6 months (resistance training ≥ 2 times/week, moderate-intensity aerobic exercise ≥ 3 times/week).
3. History of unstable cardiovascular disease, stroke, diabetes, psychiatric disorders, or other contraindications to exercise in the past 6 months.
4. Previously diagnosed with rheumatoid arthritis.
5. History of conditions affecting motor coordination, such as poliomyelitis sequelae, epilepsy, or stroke sequelae.
6. Presence of implanted medical devices due to previous fractures, heart disease, or other conditions.
7. Diagnosis of malignant tumors.
8. Unable to independently use the WeChat mini program used in this study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Extensor Strength | Week 12
  Measurement of the maximal isometric strength of the knee extensor muscles using a dynamometer. Assessed at week 12.

SECONDARY OUTCOMES:
Knee Extensor Strength | Week 6
  Same assessment as primary outcome but conducted at week 6.
Knee Flexor Strength | Weeks 6 and 12
  Measurement of the maximal isometric strength of the knee flexor muscles using a dynamometer. Assessed at weeks 6 and 12.
Grip Strength (Upper Limb Muscle Strength) | Weeks 6 and 12
  Assessment of upper limb strength via handgrip dynamometry, using the dominant hand. Recorded at weeks 6 and 12.
Timed Up and Go Test (TUGT) | Weeks 6 and 12
  A functional mobility test measuring the time (in seconds) it takes to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Evaluated at weeks 6 and 12.
6-Meter Gait Speed Test | Weeks 6 and 12
  Assessment of walking speed over a 6-meter distance, used to evaluate lower limb mobility. Performed at weeks 6 and 12.
6-Minute Walk Test (6MWT) | Weeks 6 and 12
  Measures the total distance (in meters) a participant can walk in 6 minutes to assess endurance. Conducted at weeks 6 and 12.
Appendicular Skeletal Muscle Mass Index (ASMI) | Weeks 6 and 12
  Index of appendicular skeletal muscle mass (kg/m²), measured by bioelectrical impedance analysis or DXA. Evaluated at weeks 6 and 12.
Reversal of Sarcopenia | weeks 6 and 12
  The reversal of sarcopenia will be assessed based on the AWGS criteria. Participants who no longer meet the diagnostic thresholds for low muscle mass and either low muscle strength or physical performance at week 12 will be classified as having experienced sarcopenia reversal

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MM, Study Director — Sports Medicine Center, West China Hospital, Sichuan University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (such as outcome measures and adherence scores) will be made available upon reasonable request within 12 months after study completion. Data access will be granted for academic research purposes only, subject to review and approval by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after study completion
Access Criteria: Request required, reviewed by PI
URL: https://www.wchscu.cn/index.html

REFERENCES:
- [Derived] Wang K, Peng L, You M, Shen B, Li J. Real-time multicomponent remote rehabilitation versus self-rehabilitation for sarcopenia: a randomized controlled trial protocol. J Orthop Surg Res. 2025 Jul 25;20(1):701. doi: 10.1186/s13018-025-06124-0. PMID 40713590